CLINICAL TRIAL: NCT02570711
Title: A Phase 2, Randomized, Proof-of-Concept Study of Nab-Paclitaxel/Gemcitabine Alone and in Combination With ACP-196 in Subjects With Previously Untreated Metastatic Pancreatic Cancer
Brief Title: Phase 2, Nab Paclitaxel/Gemcitabine Alone and in Combination With ACP-196 in Subjects With Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACE-ST-004
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Acalabrutinib
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — acalabrutinib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Regimen 1 (Experimental): ACP-196 and nab-paclitaxel and gemcitabine
  Interventions: Drug: ACP-196; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Regimen 2 (Experimental): Nab-paclitaxel and gemcitabine
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: ACP-196 — ACP-196 capsule
  Other Names: acalabrutinib
  Arms: Regimen 1
Drug: Nab-paclitaxel — Nab-paclitaxel infusion
  Other Names: ABRAXANE
Drug: Gemcitabine — Gemcitabine infusion
  Other Names: Gemzar

SUMMARY:
To evaluate the safety and efficacy of ACP-196 and nab paclitaxel/gemcitabine in subjects with previously untreated metastatic pancreatic cancer using standard response criteria

DETAILED DESCRIPTION:
A Phase 2, multicenter, open-label, randomized clinical trial. The study was to evaluate the efficacy and safety of ACP-196 plus nab-paclitaxel/gemcitabine compared with nab-paclitaxel/gemcitabine in subjects who have previously untreated metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* ECOG performance status of 0 or 1.
* Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas.
* No previous radiotherapy, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-FU or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.

Exclusion Criteria:

* Prior malignancy (other than pancreatic cancer), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 2 years.
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Biliary obstruction or presence of a percutaneous biliary drain. Note: Subjects with endobiliary stents may participate as long the enrollment criterion relating to serum bilirubin concentration is met.
* Breastfeeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trial, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (10):
- United States (10):
  - Ventura Clinical Trials, Ventura, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - International Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - ACP-196 and Nab-Paclitaxel and Gemcitabine: Acalabrutinib 100mg PO BID on Day 1 to 28 with Nab-Paclitaxel 125mg/m2 and Gemcitabine 1000mg/m2 on Days 1,8, and 15; cycles were repeated every 28 days.
- Arm 2 - Nab-Paclitaxel and Gemcitabine: Nab-Paclitaxel 125mg/m2 and gemcitabine 1000mg/m2 on Days 1,8, and 15; cycles repeated every 28 days.
Period: Overall Study
Arm/Group | Arm 1 - ACP-196 and Nab-Paclitaxel and Gemcitabine | Arm 2 - Nab-Paclitaxel and Gemcitabine
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — Early Termination of Study by Sponsor | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1- ACP-196 and Nab-Paclitaxel and Gemcitabine: Acalabrutinib 100mg PO BID on Days 1 to 28 with Nab-Paclitaxel 125mg/m2 and Gemcitabine 1000mg/m2 on Days 1,8, and 15; cycles were repeated every 28 days.
- Arm 2 - Nab-Paclitaxel and Gemcitabine: Nab-Paclitaxel 125mg/m2 and Gemcitabine 1000mg/m2 on Days 1,8, and 15; Cycles were repeated every 28 days.
- Total: Total of all reporting groups
Arm/Group | Arm 1- ACP-196 and Nab-Paclitaxel and Gemcitabine | Arm 2 - Nab-Paclitaxel and Gemcitabine | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3
ECOG Performance Status [Number; unit: participants] — The ECOG Scale of Performance Status is one such measurement. It describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.).
  participants
    ECOG - 0 | 0 | 1 | 1
    ECOG = 1 | 1 | 1 | 2
Subjects who have previously untreated metastatic pancreatic cancer [Count of Participants; unit: Participants] — Subjects who have previously untreated metastatic pancreatic cancer and meet all inclusion and exclusion criteria
  Participants | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) of ACP-196 plus nab-paclitaxel/gemcitabine compared with nab-paclitaxel/gemcitabine in patients with previously untreated metastatic pancreatic cancer
Time Frame: At screening, Cycle 3, and Day 1 of every other cycle afterwards (e.g., Cycle 5 Day 1). Every cycle is 28 days.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1- ACP-196 and Nab-Paclitaxel and Gemcitabine: ACP-196 and nab-paclitaxel and gemcitabine
  ACP-196: ACP-196 capsule
  Nab-paclitaxel: Nab-paclitaxel infusion
  Gemcitabine: Gemcitabine infusion
- Arm 2 - Nab-Paclitaxel and Gemcitabine: Nab-paclitaxel and gemcitabine
  Nab-paclitaxel: Nab-paclitaxel infusion
  Gemcitabine: Gemcitabine infusion
Arm/Group | Arm 1- ACP-196 and Nab-Paclitaxel and Gemcitabine | Arm 2 - Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm 1 - ACP-196 and Nab-Paclitaxel and Gemcitabine: Acalabrutinib 100mg PO BID on Days 1 to 28 with Nab-Paclitaxel 125mg/m2 and Gemcitabine 1000mg/m2 on Days 1,8, and 15; Cycles were repeated every 28 days.
- Arm 2 - Nab-Paclitaxel and Gemcitabine: Nab-Paclitaxel 125mg/m2 on Days 1,8, and 15; Cycles were repeated every 28 days.
Arm/Group | Arm 1 - ACP-196 and Nab-Paclitaxel and Gemcitabine | Arm 2 - Nab-Paclitaxel and Gemcitabine
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - ACP-196 and Nab-Paclitaxel and Gemcitabine (N=1) | Arm 2 - Nab-Paclitaxel and Gemcitabine (N=2)
Septic Shock (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - ACP-196 and Nab-Paclitaxel and Gemcitabine (N=1) | Arm 2 - Nab-Paclitaxel and Gemcitabine (N=2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Infusion Site Extravasation (General disorders) | 0 | 1
Peripheral Swelling (General disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT02570711/Prot_SAP_000.pdf